CLINICAL TRIAL: NCT00622622
Title: Phase I Study of Gemcitabine With Antiangiogenic Vaccine Therapy Using Epitope Peptide Restricted to HLA-A*2402 Derived From VEGFR2 in Patients With Unresectable, Locally Advanced, Recurrent or Metastatic Pancreatic Cancer
Brief Title: Gemcitabine With Antiangiogenic Peptide Vaccine Therapy in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Second Department of Surgery, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WPR2-0710
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I study (Experimental)
  Interventions: Biological: VEGFR2-169 and gemcitabine

INTERVENTIONS:
Biological: VEGFR2-169 and gemcitabine — Escalating doses of VEGFR2-169 will be administered by subcutaneous injection on days 1,8,15 and 22 of each 28-day treatment cycles(doses of 0.5,1.0,2.0mg/body are planned). Gemcitabine will be administered intravenously at a fixed dose of 1000mg/m2 on days 1,8 and 15. Repeated cycles of VEGFR2-169 and gemcitabine will be administered until patients develop progressive disease or unacceptable toxicity,or for maximum 2 cycles, whichever occurs first.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and immune response of different doses of VEGFR2-169 emulsified with Montanide ISA 51 in combination with gemcitabine and to determine the recommended phase II dose.

DETAILED DESCRIPTION:
Vascular endothelial growth factor receptor 2(VEGFR2) is essential target for tumor angiogenesis, and VEGFR2-169 induces specific Cytotoxic T lymphocytes (CTL) against VEGFR2 expressed targets. VEGFR2-169 shows strong anti-tumor effects restricted to HLA-A*2402 in vitro, and this peptide induces CTL from cancer patients. 60% in Japanese population have HLA-A*2402. VEGFR2-169 is suitable for clinical trial, and gemcitabine has been approved against pancreatic cancer. Gemcitabine is reported to improve immune-response, therefore synergistic effect between vaccine therapy and chemotherapy will be expected. In this clinical trial, we evaluate the safety, tolerability and immune response of different doses of VEGFR2-169 emulsified with Montanide ISA 51 in combination with gemcitabine and to determine the recommended phase II dose of peptide.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

1. locally advanced or metastatic pancreatic cancer precluding curative surgical resection and recurrent pancreatic cancer
2. measurable disease by CT scan

PATIENT CHARACTERISTICS

1. ECOG performance status 0-2
2. Life expectancy > 3 months
3. Laboratory values as follows

   * 2000/mm3 < WBC < 15000/mm3
   * Platelet count > 75000/mm3
   * Bilirubin < 3.0 mg/dl
   * Aspartate transaminase < 150 IU/L
   * Alanine transaminase < 150 IU/L
   * Creatinine < 3.0 mg/dl
4. HLA-A*2402
5. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy(woman of childbearing potential:Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Active or uncontrolled infection
4. Concurrent treatment with steroids or immunosuppressing agent
5. Prior chemotherapy of gemcitabine
6. Prior chemotherapy,radiation therapy, or immunotherapy within 4 weeks
7. Serious or nonhealing wound, ulcer, or bone fracture
8. Active or uncontrolled other malignancy
9. Ileus
10. Interstitial pneumonia
11. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11; Primary Completion 2006-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety(toxicities as assessed by NCI CTCAE version 3) | 3 months

SECONDARY OUTCOMES:
VEGFR2 peptide specific CTL induction in vitro | 3 months
DTH to VEGFR2 peptide | 3 months
Changes in levels of regulatory T cells | 3 months
Objective response rate as assessed by RECIST criteria | 1 year
Time to progression | 1 years
survival | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, MD, Study Chair — Wakayama Medical University, Second Department of Surgery
Locations (1):
- Wakayama Medical University Hospital, 811-1 Kimiidera, Wakayama, Wakayama, Japan

REFERENCES:
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316
- [Background] Li Y, Wang MN, Li H, King KD, Bassi R, Sun H, Santiago A, Hooper AT, Bohlen P, Hicklin DJ. Active immunization against the vascular endothelial growth factor receptor flk1 inhibits tumor angiogenesis and metastasis. J Exp Med. 2002 Jun 17;195(12):1575-84. doi: 10.1084/jem.20020072. PMID 12070285
- [Background] Niethammer AG, Xiang R, Becker JC, Wodrich H, Pertl U, Karsten G, Eliceiri BP, Reisfeld RA. A DNA vaccine against VEGF receptor 2 prevents effective angiogenesis and inhibits tumor growth. Nat Med. 2002 Dec;8(12):1369-75. doi: 10.1038/nm1202-794. Epub 2002 Nov 4. PMID 12415261
- [Background] Date Y, Kimura A, Kato H, Sasazuki T. DNA typing of the HLA-A gene: population study and identification of four new alleles in Japanese. Tissue Antigens. 1996 Feb;47(2):93-101. doi: 10.1111/j.1399-0039.1996.tb02520.x. PMID 8851721
- [Background] Correale P, Cusi MG, Del Vecchio MT, Aquino A, Prete SP, Tsang KY, Micheli L, Nencini C, La Placa M, Montagnani F, Terrosi C, Caraglia M, Formica V, Giorgi G, Bonmassar E, Francini G. Dendritic cell-mediated cross-presentation of antigens derived from colon carcinoma cells exposed to a highly cytotoxic multidrug regimen with gemcitabine, oxaliplatin, 5-fluorouracil, and leucovorin, elicits a powerful human antigen-specific CTL response with antitumor activity in vitro. J Immunol. 2005 Jul 15;175(2):820-8. doi: 10.4049/jimmunol.175.2.820. PMID 16002679
- [Background] Dauer M, Herten J, Bauer C, Renner F, Schad K, Schnurr M, Endres S, Eigler A. Chemosensitization of pancreatic carcinoma cells to enhance T cell-mediated cytotoxicity induced by tumor lysate-pulsed dendritic cells. J Immunother. 2005 Jul-Aug;28(4):332-42. doi: 10.1097/01.cji.0000164038.41104.f5. PMID 16000951
- [Derived] Miyazawa M, Ohsawa R, Tsunoda T, Hirono S, Kawai M, Tani M, Nakamura Y, Yamaue H. Phase I clinical trial using peptide vaccine for human vascular endothelial growth factor receptor 2 in combination with gemcitabine for patients with advanced pancreatic cancer. Cancer Sci. 2010 Feb;101(2):433-9. doi: 10.1111/j.1349-7006.2009.01416.x. Epub 2009 Oct 27. PMID 19930156